CLINICAL TRIAL: NCT05383885
Title: A Prospective Observational Study of the Perfusion Index an a Predictor of Return of Spontaneus Circulation in Out of Hospital Cardiac Arrest
Brief Title: Is the Perfusion Index an Accurate Predictor of Return of Spontaneus Circulation in Out-of-hospital Cardiac Arrest
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Other Study IDs: CE/21-11-01
Record Dates: First submitted 2022-05-03; First posted 2022-05-20 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-05

CONDITIONS: Death, Sudden, Cardiac; Perfusion Index; Return of Spontaneous Circulation
Keywords: cardiac arrest; perfusion index; Return of spontaneous circulation; End tidal CO2
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational cohort: The study is an observational study on a single cohort of consecutive out-of-hospital cardiac arrest patients.
  All patients in the cohort will be monitored with a non-invasive pletismograph. No intervention will be administered to any patient and no decision on treatment will be based on the collected informations. Treating physicians will be blinded to collected values of perfusion index during the study

SUMMARY:
The purpose of this pilot feasibility study is to evaluate the ability of the Perfusion Index to predict the return to spontaneous circulation of the out-of-hospital cardiac arrest patient during cardiopulmonary resuscitation.

The performance of the perfusion index will also be compared to the current gold standard, end-tidal CO2 (EtCO2).

DETAILED DESCRIPTION:
The aim of this observational research is to measure the predictive performance the perfusion index to predict a return of a spontaneous circulation (ROSC) during cardiopulmonary resuscitation (CPR).

The research focuses on patients in out-of-hospital cardiac arrest (OHCA) and in-hospital cardiac arrest (IHCA) treated by the mobile intensive care unit of Saint Pierre University Hospital.

The study will be a pilot observational study during cardiac arrest. During the study period a non-invasive sensor will be connected to the patient's finger to measure continously and non-invasively the perfusion index. This non-invasive measurement is done by means of an infrared light which has no known risks for the health of the patient and which is usually used for the measurement of arterial oxygen saturation (SatO2). No intervention is planned as no decision will be taken on treatment based on the collected values of perfusion index during the arrest and post-arrest care of the participants.

The study will therefore be conducted during conventional advanced life support procedures without rescuers having access to the ongoing measurements.

The study will end when the participant returns to spontaneous circulation (RACS) or when patients is admitted to the emergency ward, whichever comes first in a time frame of maximum two hours.

The decision to stop resuscitation procedures will be made in accordance with the European Resuscitation Council (ERC) recommendations and the Resuscitation Termination Rules (TOR) for cardiac arrest.

Pulsatility index values will be sampled at a 0.5 Hertz frequency. These values will be tested for their ability to predict ROSC within 2 minutes. Similarly, EtCO2 values (as a gold standard) will be analyzed from the time of first measure. The sensitivity and specificity of the collected values of EtCO2 in the prediction of ROSC will be compared, at the end of the study to the diagnostic sensibility and specificity of different thresholds of the perfusion index.

The patient's consent will be requested at the moment when he/she recovers consciousness allowing the comprehension and signature of a consent after the cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Out of hospital cardiac arrest with an indication to initiate chest compressions
* In hospital cardiac arrest with an indication to initiate chest compressions

Exclusion Criteria:

* Pregnant patients
* Prisoners

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with out-of-hospital or in-hospital cardiac arrest will be assessed for eligibility.
  After verifiying inclusion and exclusion criteria patients will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Return of Spontaneous Circulation - Perfusion index - absolute values | From study inclusion until hospital admission or date of death from any cause, whichever came first, assessed up to 2 hours after inclusion
  Receiver operating characteristic curve of the perfusion index to predict return of spontaneous circulation. Area under the curve of the receiver operating curve will be measured and reported for absolute values.
Return of Spontaneous Circulation - Perfusion index - trend values | From study inclusion until hospital admission or date of death from any cause, whichever came first, assessed up to 2 hours after inclusion
  Receiver operating characteristic curve of the perfusion index to predict return of spontaneous circulation. Area under the curve of the receiver operating curve will be measured and reported for trend values of the pulsatility index.

SECONDARY OUTCOMES:
Return of Spontaneous Circulation - EtCO2 - Perfusion index | From study inclusion until hospital admission or date of death from any cause, whichever came first, assessed up to 2 hours after inclusion
  A receiver operating characteristic curve of the perfusion index to predict return of spontaneous circulation will be plotted against a receiver operating characteristic curve of end-tidal CO2 to predict return of spontaneous circulation. Area under the curve of the two receiver operating curve will be compared and assessed for superiority.

OTHER OUTCOMES:
Re-arrest - Perfusion index | From return of spontaneous circulation until hospital admission or re-arrest from any cause, whichever came first, assessed up to 2 hours after inclusion
  Receiver operating characteristic curve of the perfusion index to predict re-arrest. Area under the curve of the receiver operating curve will be measured and reported for absolute values.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Saint Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available to other researcher as csv excell file one month after publication
Supporting Information: ICF, Analytic Code
Time Frame: One month after publication, indefinitely.
Access Criteria: Any researcher with access to figshare

DOCUMENTS (1):
  • Study Protocol (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT05383885/Prot_000.pdf